CLINICAL TRIAL: NCT00417196
Title: A Randomized, Double-blind, Placebo-controlled Study to Assess the Safety, Pharmacokinetics and Pharmacodynamics of Single Escalating Doses of Intravenous QAX576
Brief Title: Safety, Pharmacodynamic and Pharmacokinetic Effects of QAX576 in Healthy Volunteers.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CQAX576A2101
Record Dates: First submitted 2006-12-28; First posted 2006-12-29 (Estimated); Last update posted 2010-10-01 (Estimated); Status verified 2010-09

CONDITIONS: Healthy
Keywords: pharmacodynamic effects, safety, healthy subjects,; Healthy male and female subjects

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: QAX576

SUMMARY:
This study is designed to evaluate the safety, pharmacodynamic and pharmacokinetic effects of individual escalating intravenous doses of QAX576 in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects age 18 to 45 years, inclusive, and in good health as determined by past medical history, physical examination, vital signs, electrocardiogram, and laboratory tests at screening.
* Only surgically sterilized female subjects with procedure performed at least 6 months prior to screening with supportive clinical documentation are allowed to participate in this study.
* Male subjects must be using a double-barrier local contraception, i.e., spermicidal gel plus condom, for the entire duration of the study, up to Study Completion visit (i.e., refrain from fathering a child in the 4 months following last study drug administration).
* Vital signs should be within the following ranges:

Oral body temperature 35.0-37.5°C. Supine systolic blood pressure, 90-140 mm Hg. Supine diastolic blood pressure, 50-90 mm Hg. Supine pulse rate, 50-90 beats per minute (bpm).

* When blood pressure and pulse will be taken again after 3 minutes standing, there shall be no more than a 20 mm Hg drop in systolic or 10 mm Hg drop in diastolic blood pressure and increase in heart rate (>20 bpm) associated with clinical manifestation of postural hypotension.
* Body mass index (BMI) must be within the range of 18 to 28 kg/m2. Subjects must weigh between 50 and 100 kg (inclusive).

Exclusion Criteria:

* Smokers (use of tobacco products in the previous 3 months). Smokers will be who reports tobacco use or has a urine cotinine greater than 500 ng/mL.
* Use of any prescription drugs within 4 weeks prior dosing, or over-the-counter (OTC) medication (vitamins, herbal supplements, dietary supplements) within 2 weeks prior to dosing. Acetaminophen is acceptable with clinical documentation.
* Participation in any clinical investigation within 4 weeks prior to dosing or longer if required by local regulations, and for any other limitation of participation based on local regulations.
* Donation or loss of 400 mL or more of blood within 8 weeks prior to first dosing, or longer if required by local regulation.
* Significant illness within 2 weeks prior to dosing.
* A past medical history of clinically significant ECG abnormalities.
* History of autonomic dysfunction or acute or chronic bronchospastic disease (including asthma and chronic obstructive pulmonary disease, treated or not treated) or clinically significant drug allergy or history of atopic allergy (asthma, urticaria, eczematous dermatitis). A known hypersensitivity to the study drug or drugs similar to the study drug..
* History or presence of any surgical or medical condition which, in the opinion of the investigator, may jeopardize the subject in case of participation in the study, including hepatic, hematological, or immunological, disorders..
* History of clinical schistosomiasis or travel within the preceding 6 months to an area with endemic schistosomiasis, including but not limited to Southeast Asia and Northwest Africa

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2006-12; Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of single escalating doses of QAX576 as assessed by vital signs, electrocardiogram (ECG), adverse events, laboratory evaluations, up to 96 hours after drug administration, and telemetry up until 24 hours post dose

SECONDARY OUTCOMES:
Exploration of pharmacokinetics of QAX576 and its pharmacodynamic effects on interleukin 13 (IL-13) concentration data. Samples collection at pre-dose and up to 48 hours post-dose.
Assess the immunogenicity of QAX576 in healthy subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Principal Investigator — Investigator site
Locations (1):
- Novartis Investigative Site, East Hanover, New Jersey, United States